CLINICAL TRIAL: NCT01597141
Title: Psychosis: Early Detection, Intervention and Prevention
Acronym: EDIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: Columbia University (Other); Harvard University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, William McFarlane, Principal Investigator, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01MH065367-01A1 (NIH)
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Prodromal Schizophrenia; Psychotic Disorders; Severe Bipolar Disorder With Psychotic Features; Severe Major Depression With Psychotic Features
Keywords: Prodromal; Schizophrenia; Psychosis; Family psychoeducation; Assertive community treatment; Supported employment; Supported education
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-aided Assertive Community Treatment (Experimental): The experimental treatment is a combination of family psychoeducation, assertive community treatment, supported education/employment and psychotropic medication.
  Interventions: Behavioral: Family-aided Assertive Community Treatment
- Enhanced standard treatment (Active Comparator): In this arm, the subjects will receive the same psychotropic drugs, but will receive individual case management, family education and crisis intervention.
  Interventions: Behavioral: Enhanced standard treatment

INTERVENTIONS:
Behavioral: Family-aided Assertive Community Treatment — The experimental treatment is a combination of family psychoeducation, assertive community treatment, supported education/employment and psychotropic medication.
  Arms: Family-aided Assertive Community Treatment
Behavioral: Enhanced standard treatment — In this arm, the subjects will receive the same psychotropic drugs, but will receive individual case management, family education and crisis intervention
  Arms: Enhanced standard treatment

SUMMARY:
The primary aim of this application is to conduct a randomized, controlled clinical trial of a specialized mental health service delivery system specifically developed for prodromal psychotic disorders. The intervention is Family-aided Assertive Community Treatment (FACT). The goal of the treatment is prevention of psychosis and disability. This study will assess experimentally the clinical effectiveness of this new type of mental health service. Other domains of outcome include cognitive dysfunction and functional disability.

DETAILED DESCRIPTION:
The proposed study will be part of a larger program, Portland Identification and Early Referral (PIER), under foundation, NIH and Center for Mental Health Services sponsorship, that has established a population-based system of early detection for Greater Portland, Maine. Previous and present effort has educated and trained the community-at-large and all health, education and other professionals, with the result that referrals are occurring at the expected frequency. The principal strategy is to intervene early, prior to onset, in the course of the onset of psychotic disorders to arrest the development of psychotic symptoms and functional disability. The test treatment is a specialized combination of psychoeducational multifamily group and assertive community treatment.

The project will support a team of clinical staff with the ability to: a. foster detection of prodromal disorders in the Greater Portland community by general practitioners, guidance counselors, mental health professionals and the general public; b. accurately assess individuals at high risk for psychosis; c. reliably deliver an evidence-based psychosocial and, if indicated, pharmacological treatment package using standardized methodology. The research study will test, in a randomized controlled trial, the symptomatic and functional outcome of treatment in 100 subjects ages 12 to 35 identified by that system. It will allow the analysis of key social factors contributing to psychosis and their interaction with the treatment conditions and each other.

ELIGIBILITY:
Inclusion Criteria:

* Prodromal psychotic symptoms
* Age 12-35
* In catchment area (greater Portland, Maine)

Exclusion Criteria:

* Previous or current psychotic episode
* IQ less than 70
* Outside catchment area
* Toxic psychosis

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2003-05; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R McFarlane, M.D., Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

REFERENCES:
- [Background] McFarlane WR, Susser E, McCleary R, Verdi M, Lynch S, Williams D, McKeague IW. Reduction in incidence of hospitalizations for psychotic episodes through early identification and intervention. Psychiatr Serv. 2014 Oct;65(10):1194-200. doi: 10.1176/appi.ps.201300336. PMID 24632857
- [Background] Woodberry KA, McFarlane WR, Giuliano AJ, Verdi MB, Cook WL, Faraone SV, Seidman LJ. Change in neuropsychological functioning over one year in youth at clinical high risk for psychosis. Schizophr Res. 2013 May;146(1-3):87-94. doi: 10.1016/j.schres.2013.01.017. Epub 2013 Feb 22. PMID 23434505
- [Result] McFarlane WR, Cook WL, Downing D, Verdi MB, Woodberry KA, Ruff A. Portland identification and early referral: a community-based system for identifying and treating youths at high risk of psychosis. Psychiatr Serv. 2010 May;61(5):512-5. doi: 10.1176/appi.ps.61.5.512. PMID 20439374
- See also: Describes risk factors for psychosis, current scientific understanding of psychosis and means of accessing services — http://www.preventmentalillness.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Family-aided ACT: The experimental treatment is a combination of family psychoeducation, assertive community treatment, supported education/employment and psychotropic medication.
  Family-aided Assertive Community Treatment: The experimental treatment is a combination of family psychoeducation, assertive community treatment, supported education/employment and psychotropic medication.
- Enhanced Treatment: In this arm, the subjects will receive the same psychotropic drugs, but will receive individual case management, family education and crisis intervention.
  Enhanced standard treatment: In this arm, the subjects will receive the same psychotropic drugs, but will receive individual case management, family education and crisis intervention
Period: Overall Study
Arm/Group | Family-aided ACT | Enhanced Treatment
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Family-aided ACT | Enhanced Treatment | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.48 (3.07) | 16.12 (2.75) | 16.3 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 26 | 26 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0 | 4 | 4
  Non-Hispanic | 50 | 46 | 96
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Global Assessment of Functioning (GAF) [Mean (Standard Deviation); unit: units on GAF scale] — The Global Assessment of Functioning is a widely used scale based on a Likert-keyed score assigned by an interviewer or clinician, based on a scale of 0-100, with 100 being the highest level of functioning and 0 the 3 lowest.
  units on GAF scale | 40.16 (13.93) | 36.39 (10.35) | 39.7 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Onset of Psychosis
Description: Onset of psychosis is defined as an event--a new psychotic episode with loss of insight, meeting a score criterion of 6 for one month on the Scale of the Prodromal Syndrome (SOPS), in which full psychosis is defined as havng one score or 6, on a scale of 0 to 6, with 0 representing no psychotic symptoms, and 6 representing full psychosis on any of 5 dimensions of psychosis. The assessemnt is based on the Structrued Interview for the Prodromal Syndrome (SIPS), w widely used instrument for assessing risk of psychosis in adolescents and young adults.
Time Frame: From date of randomization until the date of first documented onset of psychosis, assessed up to 60 months
Measure: Number; unit: percentage of sample converting
Arm/Group | Family-aided ACT | Enhanced Treatment
Number analyzed (Participants) | 50 | 50
percentage of sample converting | 10 | 14

2. Secondary Outcome: Functioning
Description: Global Assessment of Functioning scale (GAF) at 24 months to assess functioning in symptom, role and social relationships. Global Assessment of Functioning is a widely used scale based on a Likert-keyed score assigned by an interviewer or clinician, based on a scale of 0-100, with 100 being the highest level of functioning.
Time Frame: 24 months
Population: 15 participants in the FACT arm and 16 participants in the Enhanced Standard Treatment arm were not assessed, having discontinued participation in the study.
Measure: Mean (Standard Deviation); unit: units on GAF scale
Arm/Group | Family-aided Assertive Community Treatment | Enhanced Standard Treatment
Number analyzed (Participants) | 35 | 34
units on GAF scale | 59.83 (16.38) | 54.68 (13.38)

ADVERSE EVENTS:
Arm/Group | Family-aided Assertive Community Treatment | Enhanced Standard Treatment
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family-aided Assertive Community Treatment (N=50) | Enhanced Standard Treatment (N=50)
Suicide (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No